CLINICAL TRIAL: NCT00487565
Title: LCS® PS: A Prospective, Multi-center Clinical Investigation of the LCS® Complete Posterior Stabilized Mobile-bearing Total Knee System
Brief Title: Clinical Investigation of the LCS® Complete Posterior Stabilized Mobile-bearing Total Knee System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06005; LCS:PS
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Juvenile Arthritis
Keywords: Total knee replacement; Total knee arthroplasty; Osteoarthritis; Rheumatoid or other inflammatory arthritis; Post-traumatic or juvenile arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Juvenile | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCS Complete Posterior Stabilized knee implant (Other): Total knee arthroplasty with a posterior stabilized implant
  Interventions: Device: Total knee arthroplasty

INTERVENTIONS:
Device: Total knee arthroplasty — Total knee arthroplasty using a posterior stabilized implant
  Other Names: LCS® Complete Posterior Stabilized Mobile-bearing Knee

SUMMARY:
Prospective, multi-center clinical study to evaluate the clinical outcomes of the posterior stabilized design of the LCS® Complete Mobile-bearing Total Knee System

DETAILED DESCRIPTION:
Prospective, multi-center study to evaluate the clinical outcome of posterior stabilized design of LCS® Complete Mobile-Bearing Total Knee System. No comparison group. 12 month enrollment, 12 month post-operative evaluation. Follow-up intervals: Pre-op, 3 month, 6 month, and 12 month.

ELIGIBILITY:
Inclusion Criteria:

* M/F
* 18-80
* Diagnosis of osteoarthritis, rheumatoid , post-traumatic, inflammatory, juvenile arthritis.
* Skeletally mature, sufficient bone stock to seat and support prosthesis
* Willing/able return for follow-up.
* Subject is willing and able to provide informed patient consent for participation in the study

Exclusion Criteria:

* History of recent/active joint sepsis, charcot neuropathy, psycho-social disorders, prior knee arthroplasty on affected site, metabolic disorders of calcified tissue
* Communicable diseases that may limit follow-up
* Medical-legal or workers compensation claims.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy O'Dell, EMT, CCRA, CCRC, Study Director — DePuy
Locations (3):
- United States (3):
  - Colorado Joint Replacement, Denver, Colorado
  - Joint Reconstruction Center, Pittsburgh, Pennsylvania
  - Jordan-Young Institute, Virginia Beach, Virginia

REFERENCES:
- See also: Related Info — http://www.arthritis.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2006 and February 2011, 210 subjects were recruited and enrolled at 4 clinics by orthopaedic surgeons. Recruitment was based on the inclusion and exclusion criteria in the clinical investigation plan.
Pre-assignment Details: This was a non-randomized study so all subjects that met the inclusion/exclusion criteria received the LCS Complete Posterior Stabilized implant. Consented subjects could be excluded from the trial based on results of pre-operative clinical and/or radiographic evaluations, as per the exclusion criteria in the clinical investigation plan.
Period: Overall Study
Arm/Group | LCS Complete Posterior Stabilized Knee Implant
Started | 210
Completed | 182
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | LCS Complete Posterior Stabilized Knee Implant
Number analyzed (Participants) | 210
Age Continuous [Mean (Standard Deviation); unit: participants]
  Age | 63.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 90
Region of Enrollment [Number; unit: participants]
  United States | 180
  Switzerland | 30

OUTCOME MEASURES:

1. Primary Outcome: Knee Active Flexion
Description: Active flexion is measured by how much a patient can bend their knee on their own, without assistance.
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | LCS Complete Posterior Stabilized Knee Implant
Number analyzed (Participants) | 182
degrees | 119.2 (9.9)

ADVERSE EVENTS:
Time Frame: In this study adverse events were reporting for the length of the study which was one year.
Description: There were 30 total occurrences of which 14 were unique serious adverse events that affected 28 subjects (2 subjects experienced more than 1 serious adverse event). There were 13 total occurrences of other adverse events, of which 1 unique event (above the 5% threshold) affected 11 subjects (2 subjects experienced more than 1 other adverse event).
Arm/Group | LCS Complete Posterior Stabilized Knee Implant
Serious Adverse Events (participants affected / at risk) | 28/210
Other Adverse Events (participants affected / at risk) | 11/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCS Complete Posterior Stabilized Knee Implant (N=210)
Cardiac (Cardiac disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 4 (4)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (10)
Other-Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Dehiscence Arthrotomy (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Distal Screw Failed at the Tuberocitas Osteotomy (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Loose Cement (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Polyethylene Spin Out After Fainting (Musculoskeletal and connective tissue disorders) | 1 (1)
Other- Subpatellar Crepitation (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Wound Dehiscence (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neurological (Nervous system disorders) | 3 (3)
Respiratory System (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCS Complete Posterior Stabilized Knee Implant (N=210)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less